CLINICAL TRIAL: NCT05684302
Title: The Effect of the Free-toroidal Design Lenses on the Subjective Visual Quality in the Myopic Population
Status: Completed | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY202101
Record Dates: First submitted 2022-12-24; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-12

CONDITIONS: Myopia; Refractive Errors
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The free-toroidal design lenses — Participants were asked to wear the new design lenses (the free-toroidal design lenses) for 1 week

SUMMARY:
A prospective, self-control, double-blind design was conducted in Tianjin. Two hundred participants were assigned to wear two kinds of spectacle glasses. To examine the effect of free-toroidal design and aspherical lens on the subjective visual quality among the myopic population.

DETAILED DESCRIPTION:
A prospective, self-control, double-blind design was conducted in Tianjin. Two hundred participants were assigned to wear two kinds of spectacle glasses. To examine the effect of free-toroidal design and aspherical lens on the subjective visual quality among the myopic population. The subjective visual quality of clarity and comfort were determined using a questionnaire when first wearing the glasses and after 1week.

ELIGIBILITY:
Inclusion Criteria:

* health volunteers
* their spherical refraction from -0.50 to -8.00 Diopter, with the cylinder diopter less than -3.00 Diopter
* best corrected visual acuity (BCVA)≥ 20/20 in both eyes
* stable refraction (no change greater than 0.5 Diopter within two years)

Exclusion Criteria:

* if they had Aphakic or intraocular lens eyes, had a history of trauma, active eye disease or ocular surgery, serious systemic diseases, or had a wearing history of corneal contact lenses.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Healthy myopic people between 18 and 50 years of age
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
The clarity score | baseline visit time
  The clarity score by a questionnaire,scores on the questionnaire range from 1 to 6, with higher scores being better
The comfort score | baseline visit time
  The comfort score by a questionnaire,scores on the questionnaire range from 1 to 6, with higher scores being better

SECONDARY OUTCOMES:
Accuracy of foveal and peripheral visual acuity | baseline visit time
  Accuracy of foveal and peripheral visual acuity was assessed by the eye movement tracking device

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jalie M. Modern spectacle lens design. Clin Exp Optom. 2020 Jan;103(1):3-10. doi: 10.1111/cxo.12930. Epub 2019 Jun 20. PMID 31222837
- [Background] Gannon C, Liang R. Evolving expertise for automated lens optimization. Appl Opt. 2020 Aug 1;59(22):G129-G136. doi: 10.1364/AO.391888. PMID 32749325